CLINICAL TRIAL: NCT01965301
Title: Double-blind, Placebo Controlled, Randomized Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BP1.5375 After Single Oral Administrations Ranging From 0.5 mg to 100 mg in Healthy Male Subjects (Part 1) Followed by the Assessment of the Effect of 3 Single Different BP1.5375 Oral Doses on Polysomnography in Comparison to 50 mg Diphenhydramine and Placebo in Healthy Male Subjects (Part 2).
Brief Title: First-time-in-man, to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BP1.5375
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: P12-03/BP1.5375; 2013-000697-30 (EudraCT Number)
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BP1.5375 (Experimental): Single oral administration ranging from 0.5 mg to 100 mg
  Interventions: Drug: BP1.5375 suspension; Drug: Diphenhydramine; Drug: Placebo
- Diphenhydramine (Active Comparator): Single oral dose of diphenhydramine 50mg
  Interventions: Drug: BP1.5375 suspension; Drug: Diphenhydramine; Drug: Placebo
- Placebo (Placebo Comparator): Single oral dose
  Interventions: Drug: BP1.5375 suspension; Drug: Diphenhydramine; Drug: Placebo

INTERVENTIONS:
Drug: BP1.5375 suspension — single oral dose
Drug: Diphenhydramine — single oral dose of Diphenhydramine 50mg
Drug: Placebo — Single oral dose

SUMMARY:
Phase I Single Ascending Dose (Part 1), phase IIa Proof Of Concept (Part 2)

DETAILED DESCRIPTION:
This is a single center, Double-blind, placebo controlled, randomized study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of BP1.5375 after single oral administrations ranging in healthy male subjects (Part 1) followed by the assessment of the effect of 3 single different BP1.5375 oral doses on polysomnography in comparison to 50 mg diphenhydramine and placebo in healthy male subjects (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Healthy male subjects aged between 18 and 45 years (inclusive).
* Subjects with a body weight of at least 50 kg and a body mass index (BMI) between 18.0 and 28.0 kg/m2 (both inclusive).
* Healthy subjects, based on history, physical examination, complete laboratory evaluation, and 12-lead ECG.
* Normal arterial blood pressure (BP) and pulse rate or, if abnormal, considered not clinically significant by the investigator. Normal BP to be [100-140] mmHg systolic and [45-90] mmHg diastolic. Normal pulse rate to be [40-90] bpm after 5 minutes rest in lying position.

Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Subject with a history of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurological, psychiatric, systemic, or infectious disease, or any other condition which, in the opinion of the investigator, would jeopardize the safety of the subject, or impact the validity of the study results.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Haematology, clinical chemistry, and urinalysis results deviating from the normal range to a clinically relevant extent at screening.
* Clinically significant findings on physical examination at screening.
* 12-lead electrocardiogram (ECG) with clinically relevant abnormalities in supine position at screening.
* Positive results from urine drug screen at screening.
* Veins unsuitable for i.v. puncture on either arm (e.g., veins that are difficult to locate, access or puncture, or veins with a tendency for rupture during or after puncture).
* Treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort) within 2 weeks prior to the (first) scheduled administration of study drug, except paracetamol (maximum 1 g/day).
* Treatment with another investigational drug within 3 months prior to screening or having participated in more than four investigational drug studies within 1 year prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* History or clinical evidence of any disease, and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* Have undergone surgery or have donated an amount equal or more than 500 mL blood, or 300 mL of plasma, within 3 months prior to screening.
* Positive results from any of the hepatitis serology tests (HBsAg, anti-HCV), at screening.
* Positive results from the HIV 1 or/and 2 serology at screening.
* History of allergy to diphenhydramine or antihistaminic drugs.
* Smoking more than 5 cigarettes per day.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Single Ascending Dose - safety and tolerability (Part 1) | Study period and follow up visit will be no more than 5 weeks
  To determine the clinical and biological safety and tolerability of BP1.5375 after an oral increasing single dose administration BP1.5375.
  * Physical examination : at screening and Follow-Up; a directed physical examination pre-dose and 24 hours post-dose,
  * Vital signs : at screening, on day -2, on day 1 pre-dose then 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 24 hours post dose and FU,
  * Body temperature : at screening, on day -2, on day 1 pre-dose, then 24 hours post-dose and FU,
  * Standard 12 lead ECG recording : at screening, on day -2, on day 1 pre-dose, then 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose and FU,
  * Clinical laboratory tests: at screening, on day1 pre-dose, then 24 hours post-dose and FU,
  * 48-hour 12 leads continuous ECG Holter recording from day -1 morning until dosing and from dosing until the morning of day 2.
Proof of Concept - effect on polysomnography (Part 2) | Study period and follow up visit will be no more than 9 weeks
  To determine whether an BP1.5375 single oral dose induced an effect on polysomnography in healthy male subjects compared to diphenhydramine 50 mg and matching placebo.
  Safety and tolerability :
  Monitoring for the occurrence of AEs, changes in physical examination, vital signs (body temperature, lying and standing blood pressure and heart rate), ECG, and clinical laboratory tests. Assessments will be performed at the following time points :
  * Physical examination: at screening, on days 1 and FU,
  * Vital signs: at screening, on days 1 and 2 and FU,
  * Body temperature: at screening and FU,
  * Standard 12 lead ECG recording : at screening, on days 1 and 2 morning and FU,
  * Clinical laboratory tests : at screening, on days 1 and 2 and FU.

CONTACTS AND LOCATIONS:
Overall Officials: van Gerven Joop, MD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Leiden, Netherlands